CLINICAL TRIAL: NCT04142658
Title: A Prospective, Randomized, Active (Warfarin) Controlled, Parallel-arm Clinical Trial to Determine if Participants With an On-X Aortic Valve Can be Maintained Safely and Effectively on Apixaban
Brief Title: PROACT Xa - A Trial to Determine if Participants With an On-X Aortic Valve Can be Maintained Safely on Apixaban
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Safety
Sponsor: Artivion Inc. (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONX1801.000-C
Record Dates: First submitted 2019-10-09; First posted 2019-10-29 (Actual); Results first posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Aortic Valve Disease; Aortic Valve Stenosis; Aortic Valve Failure
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis | interventions — apixaban; Warfarin

STUDY DESIGN:
Intervention Model Description: Parallel control and treatment arm at a 1:1 ratio.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Apixaban (Experimental): Apixaban 5 mg twice daily(BID) or 2.5 mg BID
  Interventions: Drug: Apixaban 5 MG; Drug: Apixaban 2.5 MG; Device: On-X Aortic Mechanical Valve
- Warfarin (Active Comparator): Patients randomized to the warfarin arm will continue warfarin in the INR range of (2.0-3.0)
  Interventions: Drug: Warfarin; Device: On-X Aortic Mechanical Valve

INTERVENTIONS:
Drug: Apixaban 5 MG — For patients that do NOT meet the following criteria
  * age ≥ 80 years
  * weight ≤ 60 kilograms
  * creatinine ≥ 1.5 mg/dL (133 micromol/L)
  Arms: Apixaban
Drug: Apixaban 2.5 MG — For patients that meet at least 2 of the following criteria
  * age ≥ 80 years
  * weight ≤ 60 kilograms
  * creatinine ≥ 1.5 mg/dL (133 micromol/L)
  Arms: Apixaban
Drug: Warfarin — Active Control Intervention
  Arms: Warfarin
Device: On-X Aortic Mechanical Valve — Inclusion Criterion: Implantation of an On-X mechanical valve in the aortic position at least 3 months (90 days) ago.
  Other Names: On-X Ascending Aortic Prosthesis (AAP)

SUMMARY:
Currently, warfarin is the only approved anticoagulation for patients with mechanical valves. The purpose of this study is to determine if participants with an On-X Prosthetic Heart Valve / On-X aortic valve can be maintained safely and effectively on apixaban. Both the On-X aortic valve and apixaban have been approved for use by the US Food and Drug Administration (FDA) but they have not been approved to be used together.

DETAILED DESCRIPTION:
There is an unmet clinical need for an alternative to warfarin, such as a direct oral anticoagulant (DOAC), as anticoagulation in participants with an aortic mechanical prosthetic valve. Some participants may be genetically hyper- or hypo-responsive to warfarin, which makes management difficult. Another small group of participants is allergic to warfarin. A much larger group of participants has difficulty maintaining warfarin control due to dietary and drug interactions. Finally, the requirement for routine blood testing makes people reluctant to take warfarin. All of these factors drive younger participants in need of aortic valve replacement (AVR) toward selection of a tissue valve instead of a mechanical valve. Despite multiple studies (randomized, matched and risk adjusted) that show that tissue valves are associated with worse outcomes, younger participants choose this type of valve to avoid warfarin. In addition, multiple clinical studies have shown valve reoperation rates are higher for tissue valves used in these younger participants. Providing an alternative to warfarin anticoagulation may lead younger participants to choose a mechanical valve with greater durability and better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age at the time of giving informed consent.
* Participants currently receiving warfarin anticoagulation and who are able to receive warfarin with a target INR 2.0 to 3.0.
* Participants are able to take low-dose aspirin at a dose of 75 -100 mg daily or have a documented contraindication to aspirin use.
* Implantation of an On-X mechanical valve in the aortic position at least 3 months (90 days) ago.
* Female participants of childbearing potential, including those who are less than 2 years post-menopausal, must agree to, and comply with using a highly effective method of birth control (eg, barrier contraceptives [condom or diaphragm with a spermicidal gel], hormonal contraceptives [implants, injectables, combination oral contraceptives, transdermal patches, or contraceptive rings], intrauterine devices or sexual abstinence) while partaking in this study. In addition, all women of childbearing potential must agree to continue to use birth control throughout the study until last study visit.
* Informed of the full nature and purpose of the study, including possible risks and side effects, given ample time and opportunity to read and understand this information, and sign and date the written informed consent before inclusion in the study.

Exclusion Criteria:

* Mechanical valve in any position other than aortic valve.
* Any cardiac surgery in the three months (90 days) prior to enrollment.
* Need to be on aspirin >100 mg daily or a P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel, or ticlopidine).
* Known hypersensitivity or other contraindication to apixaban.
* On dialysis or a creatinine clearance < 25 mL/min.
* Ischemic stroke or intracranial hemorrhage within 3 months.
* Active pathological bleeding at the time of screening for enrollment.
* Active endocarditis at the time of screening for enrollment.
* Pregnant, plan to become pregnant, or are breast feeding.
* On concomitant combined strong P-gp and CYP3A4 inducers or inhibitors.
* History of non-compliance with recommended monthly INR testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 863 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Svensson, MD, PhD, Study Chair — Steering Committee; John Alexander, MD, Study Chair — Steering Committee
Locations (62):
- United States (62):
  - Tucson Heart Center, Tucson, Arizona
  - CHI St. Vincent Heart Institute, Little Rock, Arkansas
  - Loma Linda University Medical Center, Loma Linda, California
  - Stanford University Medical Center, Palo Alto, California
  - Sharp Memorial, San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale- New Haven Hospital, New Haven, Connecticut
  - Baycare Health / Morton Plant Hospital, Clearwater, Florida
  - Shands Hospital (University of Florida Health), Gainesville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - OSF Cardiovascular Institute, Rockford, Illinois
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Maine Medical Center, Portland, Maine
  - John's Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University Medical Center, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai- St. Luke's Hospital, New York, New York
  - NewYork-Presbyterian Hospital, New York, New York
  - NewYork-Presbyterian/ Weill Cornell Medical Center, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - University of Rochester Medical Center, Rochester, New York
  - Atrium Health Carolinas Medical Center (CMC), Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Lehigh Valley Hospital Allentown, Allentown, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Shadyside, Pittsburgh, Pennsylvania
  - Avera Health / North Central Heart, Sioux Falls, South Dakota
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - William P. Clements Jr. University Hospital, Dallas, Texas
  - TCU School of Medicine, Fort Worth, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - The Heart Hospital at Baylor Plano, Plano, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Henrico Doctors' Hospital, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Swedish Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Tacoma General Hospital, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Wauwatosa, Wisconsin

REFERENCES:
- [Background] Akins CW, Miller DC, Turina MI, Kouchoukos NT, Blackstone EH, Grunkemeier GL, Takkenberg JJ, David TE, Butchart EG, Adams DH, Shahian DM, Hagl S, Mayer JE, Lytle BW; Councils of the American Association for Thoracic Surgery; Society of Thoracic Surgeons; European Assoication for Cardio-Thoracic Surgery; Ad Hoc Liaison Committee for Standardizing Definitions of Prosthetic Heart Valve Morbidity. Guidelines for reporting mortality and morbidity after cardiac valve interventions. J Thorac Cardiovasc Surg. 2008 Apr;135(4):732-8. doi: 10.1016/j.jtcvs.2007.12.002. No abstract available. PMID 18374749
- [Background] Bourguignon T, Lhommet P, El Khoury R, Candolfi P, Loardi C, Mirza A, Boulanger-Lothion J, Bouquiaux-Stablo-Duncan AL, Marchand M, Aupart M. Very long-term outcomes of the Carpentier-Edwards Perimount aortic valve in patients aged 50-65 years. Eur J Cardiothorac Surg. 2016 May;49(5):1462-8. doi: 10.1093/ejcts/ezv384. Epub 2015 Nov 2. PMID 26530269
- [Background] Chambers JB, Pomar JL, Mestres CA, Palatianos GM. Clinical event rates with the On-X bileaflet mechanical heart valve: a multicenter experience with follow-up to 12 years. J Thorac Cardiovasc Surg. 2013 Feb;145(2):420-4. doi: 10.1016/j.jtcvs.2011.12.059. Epub 2012 Feb 17. PMID 22341654
- [Background] Eikelboom JW, Connolly SJ, Brueckmann M, Granger CB, Kappetein AP, Mack MJ, Blatchford J, Devenny K, Friedman J, Guiver K, Harper R, Khder Y, Lobmeyer MT, Maas H, Voigt JU, Simoons ML, Van de Werf F; RE-ALIGN Investigators. Dabigatran versus warfarin in patients with mechanical heart valves. N Engl J Med. 2013 Sep 26;369(13):1206-14. doi: 10.1056/NEJMoa1300615. Epub 2013 Aug 31. PMID 23991661
- [Background] Glaser N, Jackson V, Holzmann MJ, Franco-Cereceda A, Sartipy U. Aortic valve replacement with mechanical vs. biological prostheses in patients aged 50-69 years. Eur Heart J. 2016 Sep 7;37(34):2658-67. doi: 10.1093/eurheartj/ehv580. Epub 2015 Nov 11. PMID 26559386
- [Background] Goldstone AB, Chiu P, Baiocchi M, Lingala B, Patrick WL, Fischbein MP, Woo YJ. Mechanical or Biologic Prostheses for Aortic-Valve and Mitral-Valve Replacement. N Engl J Med. 2017 Nov 9;377(19):1847-1857. doi: 10.1056/NEJMoa1613792. PMID 29117490
- [Background] Granger CB, Alexander JH, McMurray JJ, Lopes RD, Hylek EM, Hanna M, Al-Khalidi HR, Ansell J, Atar D, Avezum A, Bahit MC, Diaz R, Easton JD, Ezekowitz JA, Flaker G, Garcia D, Geraldes M, Gersh BJ, Golitsyn S, Goto S, Hermosillo AG, Hohnloser SH, Horowitz J, Mohan P, Jansky P, Lewis BS, Lopez-Sendon JL, Pais P, Parkhomenko A, Verheugt FW, Zhu J, Wallentin L; ARISTOTLE Committees and Investigators. Apixaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2011 Sep 15;365(11):981-92. doi: 10.1056/NEJMoa1107039. Epub 2011 Aug 27. PMID 21870978
- [Background] Head SJ, Mylotte D, Mack MJ, Piazza N, van Mieghem NM, Leon MB, Kappetein AP, Holmes DR Jr. Considerations and Recommendations for the Introduction of Objective Performance Criteria for Transcatheter Aortic Heart Valve Device Approval. Circulation. 2016 May 24;133(21):2086-93. doi: 10.1161/CIRCULATIONAHA.115.020493. PMID 27217434
- [Background] Head SJ, Celik M, Kappetein AP. Mechanical versus bioprosthetic aortic valve replacement. Eur Heart J. 2017 Jul 21;38(28):2183-2191. doi: 10.1093/eurheartj/ehx141. PMID 28444168
- [Background] IntHout J, Ioannidis JP, Borm GF. The Hartung-Knapp-Sidik-Jonkman method for random effects meta-analysis is straightforward and considerably outperforms the standard DerSimonian-Laird method. BMC Med Res Methodol. 2014 Feb 18;14:25. doi: 10.1186/1471-2288-14-25. PMID 24548571
- [Background] Samsa G, Matchar DB, Dolor RJ, Wiklund I, Hedner E, Wygant G, Hauch O, Marple CB, Edwards R. A new instrument for measuring anticoagulation-related quality of life: development and preliminary validation. Health Qual Life Outcomes. 2004 May 6;2:22. doi: 10.1186/1477-7525-2-22. PMID 15132746
- [Background] Lester PA, Coleman DM, Diaz JA, Jackson TO, Hawley AE, Mathues AR, Grant BT, Knabb RM, Ramacciotti E, Frost CE, Song Y, Wakefield TW, Myers DD Jr. Apixaban Versus Warfarin for Mechanical Heart Valve Thromboprophylaxis in a Swine Aortic Heterotopic Valve Model. Arterioscler Thromb Vasc Biol. 2017 May;37(5):942-948. doi: 10.1161/ATVBAHA.116.308649. Epub 2017 Feb 23. PMID 28232327
- [Background] McNicholas KW, Ivey TD, Metras J, Szentpetery S, Marra SW, Masters RG, Dilling EW, Slaughter MS, Mack MJ. North American multicenter experience with the On-X prosthetic heart valve. J Heart Valve Dis. 2006 Jan;15(1):73-8; discussion 79. PMID 16480015
- [Background] Palatianos GM, Laczkovics AM, Simon P, Pomar JL, Birnbaum DE, Greve HH, Haverich A. Multicentered European study on safety and effectiveness of the On-X prosthetic heart valve: intermediate follow-up. Ann Thorac Surg. 2007 Jan;83(1):40-6. doi: 10.1016/j.athoracsur.2006.08.010. PMID 17184628
- [Background] Puskas J, Gerdisch M, Nichols D, Quinn R, Anderson C, Rhenman B, Fermin L, McGrath M, Kong B, Hughes C, Sethi G, Wait M, Martin T, Graeve A; PROACT Investigators. Reduced anticoagulation after mechanical aortic valve replacement: interim results from the prospective randomized on-X valve anticoagulation clinical trial randomized Food and Drug Administration investigational device exemption trial. J Thorac Cardiovasc Surg. 2014 Apr;147(4):1202-1210; discussion 1210-1. doi: 10.1016/j.jtcvs.2014.01.004. Epub 2014 Jan 12. PMID 24512654
- [Background] Puskas JD, Gerdisch M, Nichols D, Fermin L, Rhenman B, Kapoor D, Copeland J, Quinn R, Hughes GC, Azar H, McGrath M, Wait M, Kong B, Martin T, Douville EC, Meyer S, Ye J, Jamieson WRE, Landvater L, Hagberg R, Trotter T, Armitage J, Askew J, Accola K, Levy P, Duncan D, Yanagawa B, Ely J, Graeve A; PROACT Investigators. Anticoagulation and Antiplatelet Strategies After On-X Mechanical Aortic Valve Replacement. J Am Coll Cardiol. 2018 Jun 19;71(24):2717-2726. doi: 10.1016/j.jacc.2018.03.535. PMID 29903344
- [Background] Tossios P, Reber D, Oustria M, Holland-Letz T, Germing A, Buchwald D, Laczkovics A. Single-center experience with the On-X prosthetic heart valve between 1996 and 2005. J Heart Valve Dis. 2007 Sep;16(5):551-7. PMID 17944128
- [Background] Williams MA, van Riet S. The On-X heart valve: mid-term results in a poorly anticoagulated population. J Heart Valve Dis. 2006 Jan;15(1):80-6. PMID 16480016
- [Background] Wu Y, Butchart EG, Borer JS, Yoganathan A, Grunkemeier GL. Clinical evaluation of new heart valve prostheses: update of objective performance criteria. Ann Thorac Surg. 2014 Nov;98(5):1865-74. doi: 10.1016/j.athoracsur.2014.05.006. Epub 2014 Sep 23. PMID 25258160
- [Background] Jawitz OK, Wang TY, Lopes RD, Chavez A, Boyer B, Kim H, Anstrom KJ, Becker RC, Blackstone E, Ruel M, Thourani VH, Puskas JD, Gerdisch MW, Johnston D, Capps S, Alexander JH, Svensson LG. Rationale and design of PROACT Xa: A randomized, multicenter, open-label, clinical trial to evaluate the efficacy and safety of apixaban versus warfarin in patients with a mechanical On-X Aortic Heart Valve. Am Heart J. 2020 Sep;227:91-99. doi: 10.1016/j.ahj.2020.06.014. Epub 2020 Jun 25. PMID 32693197
- [Derived] Wang TY, Svensson LG, Wen J, Vekstein A, Gerdisch M, Rao VU, Moront M, Johnston D, Lopes RD, Chavez A, Ruel M, Blackstone EH, Becker RC, Thourani V, Puskas J, Al-Khalidi HR, Cable DG, Elefteriades JA, Pochettino A, Wolfe JA, Graeve A, Sultan I, Sabe AA, Michelena HI, Alexander JH. Apixaban or Warfarin in Patients with an On-X Mechanical Aortic Valve. NEJM Evid. 2023 Jul;2(7):EVIDoa2300067. doi: 10.1056/EVIDoa2300067. Epub 2023 May 6. PMID 38320162

RESULTS

PARTICIPANT FLOW:
Groups:
- Apixaban: Apixaban 5 mg twice daily(BID) or 2.5 mg BID
  Apixaban 5 MG: For patients that do NOT meet the following criteria
  * age ≥ 80 years
  * weight ≤ 60 kilograms
  * creatinine ≥ 1.5 mg/dL (133 micromol/L)
  Apixaban 2.5 MG: For patients that meet at least 2 of the following criteria
  * age ≥ 80 years
  * weight ≤ 60 kilograms
  * creatinine ≥ 1.5 mg/dL (133 micromol/L)
  On-X Aortic Mechanical Valve: Inclusion Criterion: Implantation of an On-X mechanical valve in the aortic position at least 3 months (90 days) ago.
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 433 | 430
Completed | 418 | 400
Not Completed | 15 | 30
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 4 | 13
Not completed — Withdrawal by Subject | 9 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 433 | 430 | 863
Age, Customized [Median (Inter-Quartile Range); unit: years] | 56 [47 to 63] | 55 [47 to 63] | 56 [47 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 105 | 207
  Male | 331 | 325 | 656
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 20 | 49
  Not Hispanic or Latino | 400 | 406 | 806
  Unknown or Not Reported | 4 | 4 | 8
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 3 | 5 | 8
  Black or African American | 8 | 14 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  White | 395 | 390 | 785
  Multiracial | 2 | 0 | 2
  Other | 7 | 3 | 10
  Unknown | 17 | 13 | 30
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 29.9 [26.3 to 34.3] | 30.1 [26.3 to 35.0] | 29.9 [26.3 to 34.6]

OUTCOME MEASURES:

1. Primary Outcome: Composite of Valve Thrombosis and Valve-related Thromboembolism
Description: Valve thrombosis was defined as any thrombus, not caused by infection, attached to or near an implanted On-X valve that occluded part of the blood-flow path, interfered with valve function, or was sufficiently large to warrant treatment other than continued oral anticoagulation. Valve-related thromboembolism was defined as any thromboembolic stroke, transient ischemic attack, myocardial infarction, or arterial thromboembolism to an organ or limb that was not associated with infection or an intracardiac tumor and was definitely or possibly related to the valve.
Time Frame: through study closure, a median follow-up of 13.5 months
Population: Patient years is determined by the number of events in the Intention to Treat group (all randomized participants) divided by the amount of person-time at risk.
Measure: Number; unit: events per patient-years
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 433 | 430
events per patient-years | 20 | 6

2. Primary Outcome: Major Bleeding
Description: Major bleeding defined as any episode of internal or external bleeding that caused death, hospitalization, or permanent injury or necessitated transfusion, pericardiocentesis, or reoperation.
Time Frame: through study closure, a median follow-up of 13.5 months
Population: On treatment group
Measure: Number; unit: event
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 420 | 414
event | 17 | 21

ADVERSE EVENTS:
Time Frame: through study closure, a median follow-up of 13.5 months
Description: Events collected and reported were valve thrombosis or dysfunction, stroke or TIA, myocardial infarction, arterial thromboembolism, bleeding, hospitalization and the reason for hospitalization, death and the cause of death.
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 2/433 | 1/430
Serious Adverse Events (participants affected / at risk) | 11/433 | 18/430
Other Adverse Events (participants affected / at risk) | 16/433 | 6/430
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=433) | Warfarin (N=430)
Major Bleeding (Surgical and medical procedures) | 11 (17) | 18 (21)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=433) | Warfarin (N=430)
Valve thrombosis or Valve-related thromboembolism (Surgical and medical procedures) | 16 (20) | 6 (6) — thrombus, thromboembolic stroke, thromboembolic transient ischemic attack (TIA), thromboembolic myocardial infarction, or arterial thromboembolism to another organ or limb

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04142658/Prot_SAP_000.pdf